CLINICAL TRIAL: NCT00003731
Title: First Line Chemotherapy With Temozolomide in Recurrent Oligodendroglial Tumors, a Phase II Trial
Brief Title: Temozolomide in Treating Patients With Recurrent Oligodendroglial Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-26971; EORTC-26971
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Glioma | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients with recurrent oligodendroglial tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic activity of temozolomide as first line chemotherapy in patients with recurrent oligodendroglial tumors after radiation therapy. II. Assess the objective response and duration of response of these patients given this treatment. III. Characterize the acute side effects of temozolomide in this patient population.

OUTLINE: This is an open label, multicenter study. Patients receive oral temozolomide on days 1-5. Courses are repeated every 28 days. Treatment continues for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 15-33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven oligodendroglioma or oligoastrocytoma with at least 25% oligodendroglial elements Recurrent or progressive disease following radiotherapy At least 3 months since prior radiotherapy Measurable disease by MRI or CT scan Lesion must have a diameter of at least 1 cm No progressive neurological deficits from the present recurrence No new neurological deficits interfering with daily activities No tumor causing midline shift or brain stem compression due to which a rapid deterioration is to be expected in case of no response No signs of increased intracranial pressure No extracranial disease

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.25 times upper limit of normal (ULN) AST/ALT no greater than 2 times ULN Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine clearance at least 60 mL/min Creatinine no greater than 1.25 times ULN Neurologic: See Disease Characteristics Other: Not pregnant or nursing Fertile patients must use effective contraception No other malignant or nonmalignant diseases interfering with follow-up No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study and follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified Other: No other concurrent investigational drugs No other concurrent antitumor agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1998-12; Primary Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (24):
- Belgium (3):
  - Hopital Universitaire Erasme, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - U.Z. Gasthuisberg, Leuven
- France (6):
  - Centre Hospitalier Regional de Lille, Lille
  - CHU de la Timone, Marseille
  - CHU de Nancy - Hopital Neurologique, Nancy
  - Hopital Pasteur, Nice
  - Centre Antoine Lacassagne, Nice
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Nervenklinik Bamberg, Bamberg
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Klinikum der Universitat Regensburg, Regensburg
- Italy (2):
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (3):
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Postgraduate Medical Institute, Bratislava, Slovakia
- Switzerland (4):
  - Kantonspital Aarau, Aarau
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Western General Hospital, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Background] Kouwenhoven MC, Kros JM, French PJ, Biemond-ter Stege EM, Graveland WJ, Taphoorn MJ, Brandes AA, van den Bent MJ. 1p/19q loss within oligodendroglioma is predictive for response to first line temozolomide but not to salvage treatment. Eur J Cancer. 2006 Oct;42(15):2499-503. doi: 10.1016/j.ejca.2006.05.021. Epub 2006 Aug 17. PMID 16914310
- [Result] van den Bent MJ, Taphoorn MJ, Brandes AA, Menten J, Stupp R, Frenay M, Chinot O, Kros JM, van der Rijt CC, Vecht ChJ, Allgeier A, Gorlia T; European Organization for Research and Treatment of Cancer Brain Tumor Group. Phase II study of first-line chemotherapy with temozolomide in recurrent oligodendroglial tumors: the European Organization for Research and Treatment of Cancer Brain Tumor Group Study 26971. J Clin Oncol. 2003 Jul 1;21(13):2525-8. doi: 10.1200/JCO.2003.12.015. PMID 12829671